CLINICAL TRIAL: NCT04985305
Title: A Cluster Randomized Trial of a Complex Intervention to Encourage Deprescribing Antidepressants in Nursing Home Residents With Dementia
Brief Title: Optimization of Deprescribing Antidepressants in Nursing Home Residents With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Velux Fonden (Other); Danish College of General Practitioners (Other); Region Capital Denmark (Other)
Responsible Party: Principal Investigator, Pernille Hølmkjær, Principal Investigator, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Velux00025829
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Dementia; Deprescriptions; Antidepressive Agents; BPSD
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This trial is designed as a cluster randomized, non-blinded parallel group superiority trial with 1:1 allocation ratio. Enhanced care-as-usual will be used as a comparator.
Who Masked: Outcomes Assessor
Masking Description: The GPs are blinded to their allocation prior to recruiting patients. Due to the nature of the intervention, it will not be possible to blind the participants, providers of care or other members of the research team after the allocation. The primary outcome is blinded to the research team when analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): * Educational session for GPs
  * Instructed to complete 10-15 home visits at the nursing home with the optimizing antidepressants and other psychotropic drugs
  * Instructed to evaluate neuropsychiatric symptoms before and after the visit using a structured form
  * Instructed to complete a teaching session at the nursing home with a pre-defined teaching material
  * Instructed to contact the nursing home before the home visit to encourage participation of regular staff and relatives in the home visit or, alternatively, to obtain information from regular staff and relatives before the home visit
  * Dialogue tool
  Interventions: Behavioral: Teaching material; Behavioral: Pre-visit reflection tool; Behavioral: Dialogue tool; Behavioral: Educational session for GPs; Behavioral: Symptom assessment scale
- Control Group (Active Comparator): * Educational session for GPs
  * Instructed to complete 10-15 home visits at the nursing home with the optimizing antidepressants and other psychotropic drugs
  * Instructed to evaluate neuropsychiatric symptoms before and after the visit using a structured form
  Interventions: Behavioral: Educational session for GPs; Behavioral: Symptom assessment scale

INTERVENTIONS:
Behavioral: Teaching material — The GPs receive a power-point slide show to use at the nursing home. The slide show includes a description of BPSD symptoms, what the mechanism, effect and adverse events of antidepressants and a rationale for deprescribing.
  Arms: Intervention Group
Behavioral: Pre-visit reflection tool — The GPs receive a checklist and an email template to ensure; 1) The home visit is planned on a day where the staff at the nursing home that knows the patient best is at work. 2) The staff at the nursing home contacts the relevant relatives and informs about the home visit. 3) The symptom assessment scale is complete by the nursing home staff and returned to the GP prior to the home visit
  Arms: Intervention Group
Behavioral: Dialogue tool — The dialogue tool includes a list of questions to help the GP explore the nursing home staffs', patients' and relatives' concerns and views on deprescribing antidepressants, as well as information on when to contact the GP. The intervention has been developed during a tailoring process involving GPs, nursing home staff, interviews with patients and other experts in the field.
  Arms: Intervention Group
Behavioral: Educational session for GPs — Before randomization all participating GPs receive a ½-day course on the evaluation and treatment of neuropsychiatric symptoms that occur in patients with dementia. Elaborate information about antidepressants to this population and reasons to discontinue use. A sSpecialists in general practice, pharmacology and geriatrics/gerontopsychiatrics teaches the course. The course is mandatory for the participating GPs, but voluntary for the staff at the GPs office. The course is preferably held with actual attendance, but may be converted to an online meeting due to the COVID-19 pandemic.
Behavioral: Symptom assessment scale — An email template containing 12 screening questions from the Neuropsychiatric Inventory Nursing Home Edition is given to the GPs to distribute to the nursing home prior to the home visit and 1 month after the home visit

SUMMARY:
The effectiveness of psychotropic medication on behavioral and psychological symptoms in dementia (BPDS) is limited, while they are associated with a higher risk of morbidity and mortality. Non-pharmacological treatment of BPSD is advocated as treatment of first choice. However, many general practitioners (GPs) find it difficult to initiate deprescribing and when attempting to discontinue psychotropic drugs in nursing home residents, they can face substantial barriers both among nursing home staff and relatives. Therefore, the investigators have developed an intervention specifically aimed at increasing knowledge on deprescribing and improving communication and collaboration between GPs, nursing home staff, relatives and patients to optimize the pharmacological treatment of BPSD.

DETAILED DESCRIPTION:
It is estimated that more than 87.000 in Denmark are living with dementia, with more than 8000 new cases each year. The majority of older persons with dementia are living at home but in a minority problems with daily activities necessitates relocation to a nursing home. Besides cognitive impairment, up to 90 % of the institutionalized older people with dementia may experience behavioral and psychological symptoms of dementia (BPSD) such as anxiety, agitation, hallucinations, depression, and apathy. An overuse of antidepressants is reported and in Denmark, about half of all nursing home residents receive at least one antidepressant and many receive other psychotropic drugs such as antipsychotics, anxiolytics and hypnotics in addition to the antidepressants. However, recent research has shown that the benefits of treatment with antidepressants in patients suffering from dementia are limited while increasing the risk of falls and cardiovascular adverse events in institutionalized older persons. Given the limited effectiveness of psychotropic medication and its high risk of side-effects such as dizziness and falls, the use of antipsychotics and anxiolytics have been recommended against for a long period, while recommendations considering antidepressants have been more mixed. Danish national guidelines recommend against the use of antidepressants in older people suffering from dementia and advocate non-pharmacological treatment of BPSD as treatment of first choice.

However in contradiction with the guidelines, a recent study showed that moving into a nursing homes, was accompanied with an increase in the number of new drug treatments including antidepressants and that this number remained unchanged for at least two years. Studies on the implementation and retention of strategies to discontinuation of psychotropic medication have shown varying effects. A recent qualitative systematic review has shown that discontinuation is often hindered by 1) the GP not getting the necessary information from the staff, 2) both relatives and staff can have concerns about the reduction or discontinuation of psychotropic medication or 3) the GP does not feel sufficiently competent/confident on their knowledge of the medication to make adjustments. These factors complicate the evaluation and adjustment of pharmacological treatment of neuropsychiatric symptoms. A Danish national strategy to try to reduce antipsychotics have been initialized in 2020, but to our knowledge there is no focused initiative to reduce antidepressants.

In Denmark each patient has a General Practitioner (GP), and the majority of nursing homes in the Capital Region has a GP who is affiliated with the nursing home. The patients may choose to accept this GP as their nursing home physician when moving to the nursing home. A nursing home physician helps improve continuity and reduces the risk of hospitalization for the patients when compared to patients without a nursing home physician.

The investigators therefore chose to apply the intervention to the nursing home physicians and their patients since more and more patients are having a nursing home physician and research has shown that is reduces amongst other things, hospitalization. Since the study is a cluster randomized controlled study set place in the Capital Region of Denmark, the investigators first invited nursing home physicians to participate. In order to be included, they had to have at least 10 patients at a nursing home.

ELIGIBILITY:
Inclusion Criteria:

* ≥72 years old
* Either have a diagnosis of dementia or have a severe cognitive impairment as judged by the GP
* Are permanently living at the nursing home
* Are prescribed at least one antidepressant with the following ATC-codes

  * Selective serotonin reuptake inhibitors (SSRIs): N06AB10 (Escitalopram); N06AB04 (Citalopram); N06AB08 (Fluvoxamin); N06AB03 (Fluoxetin); N06AB05 (Paroxetin); N06AB06 (Sertralin);
  * Serotonin-Norepinephrine Reuptake inhibitors (SNRIs): N06AX21 (Duloxetin); N06AX16 (Venlafaxin);
  * Tricyclic antidepressants (TCAs): N06AA09 (Amitriptylin); N06AA04 (Clomipramin); N06AA02 (Imipramin); N06AA10 (Nortriptylin); (Dosulepin); N06AA17
  * Noradrenergic and specific serotonergic antidepressants (NaSSAs) / Atypical antidepressants N06AX03 (Mianserin); N06AX11 (Mirtazapin);
  * Monoamine oxidase inhibitors (MAOIs):N06AF01 (Isocarboxazid);
  * Noradrenaline reuptake inhibitor (NARI): N06AX18 (Reboxetin);
  * Other antidepressant with effect on the serotonin-system: N06AX26 (Vortioxetin);
  * Melatonin agonists: N06AX22 (Agomelatin);

Exclusion Criteria:

* They are under treatment of a psychiatrist.
* They are enrolled in another psychopharmacological trial
* There is a suspicion of a current clinical, major depression or suicidal behavior and intentions.
* Receiving end-of-life care

Min Age: 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Reduction of antidepressant | Intervention period of three months for each patient.
  The primary outcome is any reduction of any antidepressant from pre- to post intervention during the intervention period, in the intervention group compared to the control group, measured as a dichotomized response (reduction; yes/no). In case of reduction of an antidepressant and an addition of another antidepressant this will not be considered a reduction

SECONDARY OUTCOMES:
Change in percentage of all antidepressants | Intervention period of three months for each patient.
  A change in percentage of total amount of antidepressants per patient prescribed from pre- to post intervention
Change in percentage of each class of antidepressants | Intervention period of three months for each patient.
  A change in percentage of each class of antidepressants per patient prescribed from pre- to post intervention
Change in percentage of other psychotropic drugs | Intervention period of three months for each patient.
  A change in percentage of number of antipsychotics, anxiolytics, hypnotics, anticonvulsants, analgesics and anti-dementia drugs prescribed per patient from pre- to post intervention
Change in BPSD symptoms | 4 weeks
  Change in outcome severity of behavioural and psychological symptoms as assessed by the symptom scale 4 weeks after the home visit
Hospital admission | Intervention period of three months for each patient.
  Number of hospital admissions during the intervention period
Falls | Intervention period of three months for each patient.
  Number of falls requiring hospital admission or emergency department visit during the intervention period
Mortality | Intervention period of three months for each patient.
  Mortality at the end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Pieter Rozing, MD, Ph.D., Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, department of Public Health, section of General Practice, Copenhagen, Denmark

REFERENCES:
- [Derived] Holmkjaer P, Rozing MP, Overbeck G, Siersma V, Holm A. Effects of deprescribing antidepressants in nursing home residents with dementia-a cluster randomized controlled trial. BMC Prim Care. 2025 Jun 3;26(1):190. doi: 10.1186/s12875-025-02894-y. PMID 40462023
- [Derived] Shahrzad S, Overbeck G, Holm A, Hoj K, Holmkjaer P. Factors promoting and impeding efforts to deprescribe antidepressants among nursing home residents with dementia- a process evaluation guided by normalization process theory. BMC Nurs. 2024 Apr 28;23(1):287. doi: 10.1186/s12912-024-01932-x. PMID 38679697
- [Derived] Holmkjaer P, Holm A, Overbeck G, Rozing MP. A cluster-randomized trial of a complex intervention to encourage deprescribing antidepressants in nursing home residents with dementia: a study protocol. Trials. 2022 May 16;23(1):410. doi: 10.1186/s13063-022-06368-9. PMID 35578351